CLINICAL TRIAL: NCT03409926
Title: The Need for FibEr Addition in SympTomatic Heart Failure
Acronym: FEAST-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Justin Ezekowitz, Professor of Medicine, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00078692
Record Dates: First submitted 2018-01-18; First posted 2018-01-24 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Heart Failure
Keywords: Heart Disease; Cardiovascular Disease; Diet; Fiber; Microbiome
MeSH Terms: conditions — Heart Failure; Heart Diseases; Cardiovascular Diseases | interventions — Gum Arabic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Microcrystalline Cellulose (MCC) 10 grams/day (Active Comparator): non-fermentable active control
  Interventions: Dietary Supplement: Acacia Gum
- Acacia Gum 5 grams/day (Experimental): fermentable dietary fiber
  Interventions: Dietary Supplement: Acacia Gum
- Acacia Gum 10 grams/day (Experimental): fermentable dietary fiber
  Interventions: Dietary Supplement: Acacia Gum

INTERVENTIONS:
Dietary Supplement: Acacia Gum — dietary supplement will be added to the participant's usual diet

SUMMARY:
FEAST-HF is a single-centre clinical trial in ambulatory patients with chronic HF to evaluate whether dietary supplementation with acacia gum reduces HF-related biomarkers NT-proBNP and ST2 and how the gut microbiome responds to dietary supplementation with acacia gum. The hypotheses of this study are 1) that changes in the gut microbiome will be correlated with a reduction in NT-proBNP and ST2 in patients with HF after treatment with acacia gum, and 2) gut microbiome configurations (composition, diversity), stability and function (gene content) will be significantly altered in patients with HF in response to acacia gum.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Willing and able to provide informed consent
* Patients with established Heart Failure (as per their treating physician) including those with both reduced and preserved ejection fraction

Exclusion Criteria:

* Patients requiring a special diet that would prohibit the intervention (e.g. celiac disease, irritable bowel disease)
* Patients who do not control their own meals (e.g. meals-on-wheels, long-term care)
* Patients with conditions that would interfere with the analysis of the microbiome (e.g. chronic diarrhea, recent antibiotics within the past month)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-09-13 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
NT-proBNP | 12 weeks
  change in NT-proBNP level

SECONDARY OUTCOMES:
Composite Clinical Outcomes | 12 weeks
  All cause death, hospitalizations and emergency department visits
Quality of Life | 12 weeks
  Change in quality of life assessed by the Kansas City Cardiomyopathy Questionnaire
NYHA Functional Class | 12 weeks
  Change in NYHA class treated as a categorical variable
6-Minute Walk Test | 12 weeks
  Change in 6-Minute Walk test
Fecal Microbiome Characterization | Baseline, Week 6, Week 12
  To examine the gut microbiome in a descriptive manner and characterize predominant species and those linked to Short Chain Fatty Acid production
ST-2 | 12 weeks
  change in ST-2 level

CONTACTS AND LOCATIONS:
Overall Officials: Justin Ezekowitz, MBBCh, Principal Investigator — University of Alberta
Locations (3):
- Canada (3):
  - University of Calgary, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Mazankowski Heart Institute, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Colin-Ramirez E, Alemayehu W, McAlister FA, Howlett JG, Willing BP, Forgie A, Madsen K, Dyck JRB, Ezekowitz JA. The Need for Fiber Addition in Symptomatic Heart Failure (FEAST-HF): A Randomized Controlled Pilot Trial. CJC Open. 2023 Jul 18;5(10):760-769. doi: 10.1016/j.cjco.2023.07.005. eCollection 2023 Oct. PMID 37876886